CLINICAL TRIAL: NCT01496742
Title: A Randomized, Phase II, Multicenter, Double-Blind, Placebo-Controlled Study Evaluating the Efficacy and Safety of Metmab Vs. Placebo in Combination With Either Bevacizumab + Platinum + Paclitaxel or Pemetrexed + Platinum in Patients With Untreated Stage IIIb or IV Non-Squamous NSCLC
Brief Title: A Study of Onartuzumab (MetMAb) in Combination With Bevacizumab (Avastin) Plus Platinum And Paclitaxel or With Pemetrexed Plus Platinum in Patients With Non-Squamous Non-Small Cell Lung Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Genentech, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: GO27821; 2011-003719-42 (EudraCT Number)
Record Dates: First submitted 2011-12-19; First posted 2011-12-21 (Estimated); Last update posted 2016-09-23 (Estimated); Status verified 2016-09

CONDITIONS: Non-Squamous Non-Small Cell Lung Cancer
MeSH Terms: interventions — onartuzumab; Bevacizumab; Cisplatin; Carboplatin; Paclitaxel; Pemetrexed

ARMS (4):
- Bevacizumab+MetMAb (Experimental)
  Interventions: Drug: RO5490258; Drug: bevacizumab [Avastin]; Drug: cisplatin/carboplatin; Drug: paclitaxel
- Bevacizumab+Placebo (Active Comparator)
  Interventions: Drug: Placebo; Drug: bevacizumab [Avastin]; Drug: cisplatin/carboplatin; Drug: paclitaxel
- Pemetrexed+MetMAb (Experimental)
  Interventions: Drug: RO5490258; Drug: cisplatin/carboplatin; Drug: pemetrexed
- Pemetrexed+Placebo (Active Comparator)
  Interventions: Drug: Placebo; Drug: cisplatin/carboplatin; Drug: pemetrexed

INTERVENTIONS:
Drug: Placebo — Matching RO5490258 (MetMAb) placebo iv, Day 1 of each 21-day cycle
  Arms: Bevacizumab+Placebo; Pemetrexed+Placebo
Drug: RO5490258 — 15 mg/kg iv, Day 1 of each 21-day cycle
  Other Names: MetMAb
  Arms: Bevacizumab+MetMAb; Pemetrexed+MetMAb
Drug: bevacizumab [Avastin] — 15 mg/kg iv, Day 1 of each 21-day cycle
  Arms: Bevacizumab+MetMAb; Bevacizumab+Placebo
Drug: cisplatin/carboplatin — standard dose iv, Day 1 of each 21-day cycle, 4 cycles
Drug: paclitaxel — 200 mg/m2 iv, Day 1 of each 21-day cycle, 4 cycles
  Arms: Bevacizumab+MetMAb; Bevacizumab+Placebo
Drug: pemetrexed — 500 mg/m2, Day 1 of each 21-day cycle
  Arms: Pemetrexed+MetMAb; Pemetrexed+Placebo

SUMMARY:
This multicenter, randomized, double-blind, placebo-controlled study will evaluate the efficacy and safety of RO5490258 (MetMab) in combination with either of two backbone chemotherapy regimens in the first-line setting in patients with incurable Stage IIIB or IV non-squamous non-small cell lung cancer. In Cohort 1, patients will be randomized to receive 4 cycles of bevacizumab (Avastin) 15 mg/kg iv, paclitaxel 200 mg/m2 iv, platinum (cisplatin/carboplatin) iv plus either MetMab 15 mg/kg iv or placebo on Day 1 of each 21-day cycle. In Cohort 2, patients will be randomized to receive pemetrexed 500 mg/m2 iv, platinum (cisplatin/carboplatin) iv plus either MetMAb 15 mg/m2 iv or placebo on Day 1 of each 21-day cycle. Patients who have not progressed after 4 cycles will be offered maintenance therapy with their assigned treatment of bevacizumab plus either MetMAb or placebo (Cohort 1) or pemetrexed plus either MetMAb or placebo (Cohort 2). Anticipated time on study treatment is until disease progression or unacceptable toxicity occurs.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients, >/= 18 years of age
* Histologically or cytologically confirmed Stage IIIB or Stage IV non-squamous non-small cell lung cancer (NSCLC)
* Eastern Cooperative Oncology Group (ECOG) performance status 0 or 1
* For patients who received prior adjuvant chemotherapy or chemoradiotherapy: a treatment-free interval of at least 12 months since last chemotherapy or chemoradiotherapy cycle
* Adequate tissue for central immunohistochemical (IHC) assay of Met receptor, and epidermal growth factor receptor (EGFR) testing if EGFR status is unknown
* Radiographic evidence of disease

Exclusion Criteria:

* Prior systemic treatment for Stage IIIB or IV non-squamous NSCLC
* Evidence of mixed NSCLC with a predominance of the squamous cell type
* Prior exposure to experimental treatment targeting either the hepatocyte growth factor (HGF) or Met pathway
* Patients with tumors confirmed to have EGFR-activating mutations who are suitable for anti-EGFR therapy (e.g. gefitinib or erlotinib), as determined by the investigator, unless that treatment is unavailable or refused by the patient
* Known central nervous system (CNS) disease, other than stable, treated brain metastases
* History of another malignancy in the previous 3 years, except for history of in situ cancer that was treated surgically with curative intent, localized prostate cancer that has been treated surgically with curative intent, or basal or squamous cell skin cancer
* Uncontrolled diabetes
* Pregnant or lactating women
* Impaired bone marrow, liver or renal function (as defined by protocol)
* Significant history of cardiovascular disease
* Positive for HIV infection

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 259 (Actual)
Dates: Start 2012-04; Primary Completion 2015-11 (Actual); Study Completion 2015-11 (Actual)

PRIMARY OUTCOMES:
Progression-free survival (tumor assessments according to RECIST criteria) | up to approximately 23 months
Progression-free survival: Subgroup of patients with Met diagnostic positive tumors | up to approximately 23 months

SECONDARY OUTCOMES:
Overall survival | up to approximately 23 months
Overall response rate (tumor assessments according to RECIST criteria) | up to approximately 23 months
Duration of response (time from first documented objective response to disease progression) | up to approximately 23 months
Disease control rate (rate of partial response plus complete response plus stable disease for at least 6 weeks) | up to approximately 23 months
Safety: Incidence of adverse events | up to approximately 23 months
Pharmacokinetics: serum concentration (Cmin/Cmax) | Pre- and post-dose on Day 1 of Cycles 1, 2 and 4 and at study termination
Serum concentrations of bevacizumab/paclitaxel/pemetrexed/platinum in combination with MetMAb | Pre- and post-dose on Day 1 of Cycles 1 and 4
Serum levels of anti-therapeutic antibodies (MetMAb ATAs) | Pre-dose Day 1 of Cycles 1, 2 and 4

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Genentech, Inc.
Locations (80):
- United States (30):
  - Huntsville, Alabama
  - Scottsdale, Arizona
  - Bakersfield, California
  - Fullerton, California
  - Los Angeles, California
  - Northridge, California
  - San Luis Obispo, California
  - Santa Barbara, California
  - Stanford, California
  - Grand Junction, Colorado
  - Boynton Beach, Florida
  - Hollywood, Florida
  - Orlando, Florida
  - Lawrenceville, Georgia
  - Marietta, Georgia
  - Harvey, Illinois
  - Fort Wayne, Indiana
  - Indianapolis, Indiana
  - Muncie, Indiana
  - Metairie, Louisiana
  - Minneapolis, Minnesota
  - Las Vegas, Nevada
  - New York, New York
  - Hickory, North Carolina
  - Cleveland, Ohio
  - Columbus, Ohio
  - Middletown, Ohio
  - Bend, Oregon
  - Portland, Oregon
  - Seattle, Washington
- Argentina (3):
  - Buenos Aires
  - La Rioja
  - Santa Rosa
- France (3):
  - Grenoble
  - Paris
  - Rennes
- Germany (5):
  - Göttingen
  - Halle
  - Immenhausen
  - München
  - Münster
- Israel (5):
  - Afula
  - Ashkelon
  - Holon
  - Tel Aviv
  - Ẕerifin
- Italy (6):
  - Avellino, Campania
  - Udine, Friuli Venezia Giulia
  - Rome, Lazio
  - Cremona, Lombardy
  - Milan, Lombardy
  - Orbassano, Piedmont
- Latvia (3):
  - Daugavpils
  - Liepāja
  - Riga
- Malaysia (5):
  - George Town
  - Kuala Lumpur
  - Negeri Sembilan
  - Pulau Pinang
  - Tanjung Bungah
- Mexico (3):
  - Aguascalientes
  - Chihuahua City
  - León
- Philippines (4):
  - Cebu City
  - Davao City
  - Pasig
  - Quezon City
- Spain (4):
  - Barcelona, Barcelona
  - Madrid, Madrid
  - Pamplona, Navarre
  - Zaragoza, Zaragoza
- Taiwan (4):
  - Kaohsiung City
  - Taichung
  - Tainan
  - Taipei
- United Kingdom (5):
  - Aberdeen
  - Birmingham
  - Bournemouth
  - Leeds
  - Manchester